CLINICAL TRIAL: NCT06931392
Title: Expectations and Experiences With Virtual Reality Training Among ICU Physicians and Nurses
Acronym: ExpertVR-ICU
Status: Not yet recruiting | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Tereza Prokopova, MD, MD, PhD, Brno University Hospital
Other Study IDs: ExpertVR-ICU
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Virtual Reality; Education; Intensive Care Unit ICU
Keywords: virtual reality; education; intensive care unit; training; European survey; physicians; nurses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to describe the expectations and experiences with virtual reality in physicians and nurses working in the European ICUs. The main questions it aims to answer are:

What emotions and worries does the expected training with virtual reality evoke? What are the potential factors causing negative emotions and fear from expected training? What is the institutional approach to the online training approach regarding participation in working hours and covering the costs? How does the experience of training using virtual reality spread among the population of ICU physicians and nurses? Participants will fill out an electronic survey.

DETAILED DESCRIPTION:
The need for constant training envelopes every medical speciality. Anesthesiology and Intensive Care or Critical care are no exceptions. Virtual reality is a very modern and fast-growing field with huge potential for education and training. The investigators hypothesise that virtual reality and online education could improve healthcare professionals' education feasibility. The survey was developed based on a trial version carried out only in the Czech Republic on 120 participants without any comments about questions clarity. The questionnaire contains a descriptive part and an explorative part about expectations and experiences with virtual reality in training. The study will aim for European ICUs. After that, the responses will be interpreted using statistical methods that fit. The investigators aim to publish our findings in a journal in WoS.

ELIGIBILITY:
Inclusion Criteria:

* HCPs working in ICU.

Exclusion Criteria:

* HCPs not working in ICU.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians and nurses working in ICU.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
What emotions and worries does the expected training with virtual reality evoke? | 6 months
  This survey is going to explore the emotions that are provoked by training in virtual reality.
What are the potential factors causing negative emotions and fear from expected training? | 6 months
  This survey describes the potential factors causing negative emotions evoked by virtual reality training.

SECONDARY OUTCOMES:
What is the institutional approach to the online training approach regarding participation in working hours and covering the costs? | 6 months
  This study explores the institution's approach to online training. Mostly in are areas of fee cover and participation during working hours.
How is the experience of training using virtual reality spread among the population of ICU physicians and nurses? | 6 months
  This study explores the experience of ICU physicians and nurses with training with virtual reality elements.

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be available on request to primary investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 1 year
Access Criteria: On request. Contact person primary investigator.